CLINICAL TRIAL: NCT07279844
Title: An Open-label, Observational, Long-term Follow-up Study Evaluating the Safety and Efficacy of RGL-193 Putamen Injection in Patients With Primary Parkinson's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: RGL-193-LTS
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum, Vector
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects who have previously participated in RGL-193-related studies and have received RGL-193 treat
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Long-term observational

SUMMARY:
To evaluate the long-term safety of RGL-193 capsid injection in patients with primary Parkinson's disease over 5 years

DETAILED DESCRIPTION:
An open-label, observational, long-term follow-up study evaluating the safety and efficacy of RGL-193 capsid injection in patients with primary Parkinson's disease over 5 years

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have previously participated in RGL-193-related studies and have received RGL-193 treatment；
2. Those who voluntarily participate in this trial and sign a written informed consent form -

Exclusion Criteria:

None

-

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mid-to-late stage Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2029-12-14 (Estimated); Study Completion 2029-12-14 (Estimated)

PRIMARY OUTCOMES:
To evaluate the long-term safety of RGL-193 capsid injection in patients with primary Parkinson's disease over 5 years | 52 weeks after core-shell injection

SECONDARY OUTCOMES:
Assess the metabolic activity of related enzymes in patients with primary PD over 5 years following RGL-193 capsid injection. | 52 weeks after core-shell injection

CONTACTS AND LOCATIONS:
Overall Officials: Chaoshi Niu, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China

IPD SHARING:
Plan to Share IPD: Undecided